CLINICAL TRIAL: NCT02357953
Title: Measurement of Cardiac Index by Transpulmonary Thermodilution Using an Implanted Central Venous Access Port: a Prospective Study in Patients Scheduled for Oncologic High-risk Surgery
Brief Title: Transpulmonary Thermodilution Using an Implented Central Venous Access Port
Acronym: ThermoD-PAC
Status: Completed | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A00003-40; 2012/1386 (Other: CSET number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Medical Oncology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measurement of cardiac index

SUMMARY:
Perioperative hemodynamic optimization requires monitoring adapted to the risks of the surgery and the patient. The investigators currently use a local hemodynamic protocol based on the data of the literature. According to this protocol, specific patients may require cardiac index and central venous oxygen saturation monitoring. the investigators chose to monitor the cardiac index (CI) with the transpulmonary thermodilution technique (TPTD) (PiCCO, Pulsion Medical System, Munich, Allemagne). The technique is based on the injection of a cooled bolus of saline into a central vein with a central venous catheter (CVC). The variation of temperature is measured with an arterial femoral catheter and allows the assessment of the cardiac output according to Stewart-Hamilton's theory. Many studies showed the reliability of this technique (Bein J Cardio Thorac Vasc Anesth 2004, Buhre Cardio thorac vasc anesth 1999, Felbinger J Clin ANesth 2005, Felbinger TW J Clin Anetsh 2002, Godie O Ann Thorac Surg 1999).

In our institute, most of the patients are fitted with a port for chemotherapy or parenteral nutrition. When PiCCO monitoring is necessary, a central venous catheter is inserted on the opposite side of the permanent implantable venous port. Indeed, insertion of the CVC can be more difficult because of the port. It may be interesting to use the port for TPTD in order to avoid the insertion of a new CVC. This would be possible only if the measurement of CI by the port was as reliable as the classical measurement with a CVC.

The aim of this study was to assess whether measurement of the CI by TPTD was possible and reliable via the port. The investigators conducted a prospective study comparing the measurement of the CI by TPTD before and after fluid challenge via the port versus the CVC.

ELIGIBILITY:
Inclusion Criteria:

* presence of port
* scheduled surgery with perioperative optimization requirement according to the local hemodynamic protocol
* oral consent of the patient after oral and written information

Exclusion Criteria:

* age inferior to 18
* Contraindication or failure to the insertion of the CVC
* Contraindication to the use of the port : local or general infection suspected or proved, absence of blood backflow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for onoclogic hish-risk surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the measurement of cardiac index with the transpulmonary thermodilution technique | At inclusion
  During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Eghiain, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France